CLINICAL TRIAL: NCT04615663
Title: Assessment of Personal, Psychosocial, Work, and Economic Burden in Patients With Mast Cell Disorders,
Brief Title: Assessment of Burden Disease in Patients With Mast Cell Disorders
Acronym: MCD&BuDi
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0354
Record Dates: First submitted 2020-06-16; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Mastocytosis; Cutaneous
Keywords: Burden; quality of life; mast cell disease; work impairment
MeSH Terms: conditions — Mastocytosis; Mast Cell Activation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- face-to-face patients: During this visit, the investigator will complete the SMI score.
  Interventions: Behavioral: Score SMI
- Email patients: this visit at M0 + 7d will correspond to the emailing of the Mc_QoL and Burden_MCD questionnaires completed by the patient.

INTERVENTIONS:
Behavioral: Score SMI — the investigator will complete the SMI score
  Groups: face-to-face patients

SUMMARY:
The symptoms caused by mast cell disorders can have a significant impact on the state of health of individuals, constituting a real burden for them, and consequently altering their quality of life. It therefore seems important to clarify the impact on the quality of life, on the psycho-affective sphere, on professional life and on the direct and indirect costs caused by the disease, as well as on the "patient's remaining burden". It seems possible by a longitudinal study (patient follow-up over 1 year).

Primary objective is Assessment of quality of life in adult patient with mast cell diseases at M0.

DETAILED DESCRIPTION:
Mast cell activation symptoms are due to the release of mast cell mediators after uncontrolled activation of mast cells. The release by mast cells of mast cell mediators (tryptase, histamine, prostaglandins, serotonin) results in mast cell activation symptoms, found in mast cell activation syndrome but also in mastocytosis. These symptoms interested the skin, gastrointestinal gut, pulmonary, cardiovascular and neuropsychiatric organs, etc.

In mastocytosis, along with these symptoms of mast cell activation, the infiltration of different organs by abnormal mast cells produces many clinical signs related to the excess of monoclonal mast cells present in the organs.

According to our clinical experience, the impact of mast cell disorder on various dimensions of life, including economic life, seems important, but it has never accurately evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years old) with confirmed mast cell disorder according to international criteria
* Patient affiliated to social security regime

Exclusion Criteria:

* Patient under legal protection (guardianship, curators or court order)
* Patient does not speak French

Ages: 18 Months to 65 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Prospective, descriptive study, both transversal and longitudinal, open, monocentric, performed in 200 patients with mast cell disease and follow-up at the CEREMAST Toulouse
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-28 (Actual); Primary Completion 2021-01-28 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Quality of life of mast cell disorder patients | Baseline
  Quality of life is evaluated with the WHOQOL-bref questionary. This validated questionnaire in French assesses six dimensions of quality of life.

SECONDARY OUTCOMES:
Mast cell disorder patient's life quality | 6 months
  Quality of life is evaluated with the WHOQOL-bref.
Mast cell disorder patient's quality of life | 12 months
  Quality of life is evaluated with the WHOQOL-bref.

CONTACTS AND LOCATIONS:
Overall Officials: LIVIDEANU Cristina, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Cristina BULAI LIVIDEANU, Toulouse, France